CLINICAL TRIAL: NCT06919068
Title: Colonic Capsule Endoscopy for Screening of Neoplasms in Patients With Anaerobic Bacteremia
Brief Title: Examination of the Large Intestine With Camera Capsule in Patients With Blood Stream Infection With Gut-associated Bacteria
Acronym: AB-care
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VEK_ID_S-20240090
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (CRC); Colorectal Cancer and Pre-cancer Polyps; Blood Stream Infection; Anaerobic Infection; Bacteriaemia
Keywords: Colorectal Cancer; Anaerobic bacteria; Bacteria, anaerobic; Cancer, colorectal; Bacteremia; Blood stream infection; Colon capsule endoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Bacteremia | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Colon capsule endoscopy — PillCam Colon 2

SUMMARY:
The goal of this observational study is to diagnose colorectal cancer or precancerous tumors in participants over the age of 18 hospitalized with blood stream infection with anaerobic gut-associated bacteria. The main question it aims to answer is:

• How prevalent is cancer and precancerous tumors in the large intestines and rectum in patients with anaerobic bacteremia? Participants will be offered an examination using colon capsule endoscopy 4-8 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Blood culture with growth of one or more of the following bacterial genera Bacteroides, Clostridium, Filifactor, Fusobacterium, Gemella, Granulicatella, Parvimonas, Peptostreptococcus, Prevotella, Solobacterium, Peptoniphilus, Ruminococcus, Finegoldia and Streptococcus.
* Able to provide oral and written informed consent
* Able to read and speak Danish

Exclusion Criteria:

* Prior colorectal cancer diagnosis
* History of stenosis of the gastrointestinal tract
* Previous treatment of inflammatory bowel disease
* Previous major surgery of the gastrointesinal tract (e.g. gastric bypass)
* Colostomy
* Pacemaker/ICD
* Pregnancy or breastfeeding
* Allergies to the bowel preparation regimen
* Severe kidney disease
* Focus of infection in skin and soft tissue or outside the truncus (e.g. decubitus, diabetic foot ulcer)
* Tumor in the colon or rectum at diagnostic imaging
* Transfer to other hospital outside the region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Odense University Hospital with anaerobic blood stream infection.
  Patients who are discharged before result of blood culture with anaerobic gut-associated bacteria, will be contacted by letter and offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer and precancerous tumors | 4-8 weeks after hospitalization with anaerobic gut-associated bacteria
  Prevalence of colorectal cancer and precancerous tumors using colon capsule endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laupland KB, Edwards F, Furuya-Kanamori L, Paterson DL, Harris PNA. Bloodstream Infection and Colorectal Cancer Risk in Queensland Australia, 2000-2019. Am J Med. 2023 Sep;136(9):896-901. doi: 10.1016/j.amjmed.2023.05.003. Epub 2023 May 23. PMID 37230400
- [Background] Justesen US, Nielsen SL, Jensen TG, Dessau RB, Moller JK, Coia JE, Andersen SL, Pedersen C, Gradel KO. Bacteremia With Anaerobic Bacteria and Association With Colorectal Cancer: A Population-based Cohort Study. Clin Infect Dis. 2022 Nov 14;75(10):1747-1753. doi: 10.1093/cid/ciac259. PMID 35380653
- [Background] Justesen US, Ellebaek MB, Qvist N, Iachina M, Frimodt-Moller N, Soes LM, Skovgaard S, Lemming L, Samulioniene J, Andersen SL, Dessau RB, Moller JK, Coia JE, Gradel KO. Colorectal cancer and association with anaerobic bacteraemia: A Danish nationwide population-based cohort study. J Infect. 2024 Aug;89(2):106212. doi: 10.1016/j.jinf.2024.106212. Epub 2024 Jul 2. PMID 38960102